CLINICAL TRIAL: NCT05817591
Title: Response Profiles to High-concentration Capsaicin Desensitization in Patients with Peripheral Neuropathic Pain with or Without Allodynia: a Regional Multicenter Prospective Cohort
Acronym: CAPSICAURA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Other Study IDs: 19-50
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Neuropathic Pain
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with peripheral neuropathic pain and having an indication of capsaicin patches: All patients will receive as part of routine care:
  * Three consecutive patches of 8% capsaicin in localized application for 30 to 60 minutes once every 3 months : at M0 (study inclusion), M3 and M6, or until pain scale < 4/10 (between 0 and 10),
  * Pain assessment every 1.5 months (+/-7 days), to evaluate clinical response,
  * 8% capsaicin patches if the pain assessment rises again to pain scale > 4/10, after an initial response to treatment
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — In current practice, capsaicin patch treatment is offered to patients with a 24-hour average pain level measured by the EN numerical scale : EN scale is > 4 Pain monitoring questionnaires will be completed by patients every 6 weeks : Neuropathic Pain Symptom Invetory (NPSI Score), Patients' Global Impression of Change (PGIC scale), Numerical pain scale

SUMMARY:
Prospective multicenter cohort to determine patient profiles (associated factors, including allodynia) with a better response to pain desensitization by capsaicin delivered in the form of a high concentration patch (8%), in a population of patients with peripheral neuropathic pain and followed up in a pain consultation in the Auvergne Rhône Alpes region.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age on the day of inclusion
* Patient who has been informed and has not expressed opposition to participating in the study,
* Patient with peripheral neuropathic pain (whatever the etiology), defined by :

  * "Neuropathic Pain 4" score ("DN4" score) ≥ 4/10
  * AND pain according to the numerical scale (EN) > 4/10,
  * AND stable analgesic treatment for at least 1 month,
  * AND with or without mechanical allodynia according to the Quantitative Sensory Testing (QST) : Brush test (dynamic), Von Frey test (static)
  * AND with or without thermal allodynia to hot or cold as determined by a ROLLTEMP-II® (Rolltemp is a device designed for quick screening of temperature sensibility over large body areas).
* Patient responding to an indication of desensitization to high concentration capsaicin concentration and not presenting any contra-indication.
* Patient naïve of high concentration of Capsaicin on the concerned zone
* Patient understanding French

Non-inclusion Criteria:

* Patient with pain related to complex regional pain syndrome (criteria not meeting the indication for capsaicin)
* Patient with active cancer (underlying disease and treatments may modify pain perception),
* Patient receiving or having received in the last 3 months Botulinum toxin A on the concerned area (this treatment of neuropathic pain may modulate the effect of capsaicin and disturb the demonstration of causality),
* Patient with planned surgery within the next 12 months on the painful site (surgery may cause neuropathic damage and/or bias the pain assessment),
* Patient included in an interventional research protocol,
* Patient under guardianship or curators,
* Patient under legal protection

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are identified during consultations for the treatment of their pain, carried out in the Chronic Pain Structures of the Auvergne Rhône-Alpes region. These patients must present peripheral neuropathic pain, whatever the etiology, and validated by a DN4 score ≥ 4/10 and a pain scale > 4/10, with a stable analgesic treatment for at least one month and for whom the investigator proposes a desensitization to high concentration Capsaicin.
  Inclusion of consecutive patients in a consultation/day hospitalization setting.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Factors (profiles) associated with a better initial response to pain desensitization by capsaicin | 12 months
  A patient is a responder if he has a reduction in pain, as measured by a numerical pain scale, of at least 30% from baseline. The scale used is "EN - échelle numérique" in french, "NRS - Numerical Rating Scale" in english, between 0 and 10 (0 being the absence of pain and 10 the most intense pain).

SECONDARY OUTCOMES:
Proportion [95% Confidence Interval (CI)] of patients "responder at 30%" at 1.5 months after each consecutive patch (e.g. at M4.5 for a second patch applied at M3) | 1.5 months after each consecutive patch
Proportion [95% CI] of patients "initial responder" at 50% | 12 months
Distribution of Neuropathic Pain Symptom Inventory (NPSI) score values over time: at inclusion, 3 months, 6 months, 9 months,12 months, and between inclusion and the end of follow-up | Each 3 months and over 12 months
  The NPSI scale is composed of 12 questions (10 descriptive questions of symptoms and 2 to evaluate the frequency and duration of pain). The score for the descriptive questions is between 0 and 100 (0 being the absence of pain and 10 the most intense pain).
Distribution of NPSI subscores values (Q8, Q9, Q10) over time: at inclusion, 3 months, 6 months, 9 months,12 months, and between inclusion and the end of follow-up | Each 3 months and over 12 months
Distribution of Patients' Global Impression of Change (PGIC) scale score values over time: at 1.5 months, 3 months, 4.5 months, 6 months, 7.5 months, 9 months,10.5 months, 12 months, and between inclusion and the end of follow-up | Each 1.5 months and over 12 months
  The Patients' Global Impression of Change (PGIC) scale describe the change (if any) in activity limitations, symptoms, emotions, and overall quality of life. It is between 1 and 7 (1 being no change or conditions has got worse, and 7 is a great deal better and a considerable improvement that as made all the difference).
In the subpopulation of patients with allodynia (dynamic mechanical or static or thermal): proportion [95% CI] of "responders" at 7.5 months | 7.5 months
In the subpopulation of initial responders at the 30% threshold: proportion [95% CI] of patients relapsing at 12 months, defined as pain scale (EN) > 4/10, indicating a new capsaicin patch | 12 months
Number of new initiation of analgesic treatment, defined by the addition of a molecule to the treatment given at the time of application of the first capsaicin patch | 12 months
Number of reduction of analgesic treatment, defined by the stop of a molecule compared to the treatment given at the time of the application of the first capsaicin patch | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane FERRANDO, Doctor, Principal Investigator — Centre Hospitalier Annecy Genevois
Locations (10):
- France (10):
  - Centre Hospitalier Annecy Genevois, Annecy
  - Hospices Civils de Lyon, Hôpital Pierre Wertheimer, Bron
  - Centre Hospitalier Métropole Savoie, Chambéry
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Universitaire Grenoble-Alpes, Grenoble
  - Hospices Civils de Lyon, Hôpital de la Croix Rousse, Lyon
  - Centre Léon Bérard, Lyon
  - Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne
  - Clinique Mutualiste Chirurgicale de Saint Etienne, Saint-Etienne
  - Médipôle Lyon Villeurbanne, Villeurbanne